CLINICAL TRIAL: NCT05948800
Title: Effect of Isotonic Seawater Solution on Nasal Patency in Athletes: an Interventional Randomized Prospective Cohort Study
Brief Title: Impact of Nasal Isotonic Solution Irigation on Healthy Athletes' Nasal Flow and Nasal Obstruction Exercise Outcomes
Acronym: ISOtastic!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Collaborators: Jadran Galenski laboratorij d.d. (Industry)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Assistant Professor, University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP 25I-29-II13-23-03
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Nasal Obstruction; Nasal Disease
Keywords: nasal irrigation; isotonic solution; NOSE questionnaire; Peak Inspiratory Nasal Flow; Excercise
MeSH Terms: conditions — Nasal Obstruction; Nose Diseases | interventions — Nasal Lavage

STUDY DESIGN:
Intervention Model Description: The participants will be divided into two groups using the binary coin-toss method (random.org) with similar physical and demographic characteristics. The first group will use an isotonic seawater solution as a nasal spray for 10 days, while the control group will not use such a solution. The group with the isotonic seawater solution applied as a nasal spray will use it at least three times a day, and necessarily before exercise (about 20 minutes before).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spraying group (Experimental): The first group will use an isotonic seawater solution as a nasal spray for 10 days. The group with the isotonic seawater solution applied as a nasal spray will use it at least three times a day, and necessarily before exercise (about 20 minutes before).
  Interventions: Dietary Supplement: Nasal irrigation with seawater isotonic solution
- Non-spraying group (No Intervention): The control group will not use such a solution.

INTERVENTIONS:
Dietary Supplement: Nasal irrigation with seawater isotonic solution — Isotonic sea water: product from the market, Aqua Maris nasal spray (manufacturer JGL, Rijeka), applied in accordance with the approved Instructions for Consumers.
  Arms: Spraying group

SUMMARY:
Nasal patency is an important component of performing exercises because it helps in humidifying, heating and filtering the inhaled air. However, many athletes and exercisers experience difficulty breathing through their nose, which can affect their breathing and performance. Namely, during sports activities and greater physical effort, there is increased air flow, which causes significant dehydration and cooling of the mucous membrane of the upper respiratory system. This dehydration is associated with the release of inflammatory mediators, which can ultimately lead to narrowing of the airways (eg in athletes with asthma). However, in all athletes, regardless of whether they have asthma or not, damage to the airways can occur because during exercise, hyperpnea exposes the respiratory epithelium to increased physical forces and pressure, which leads to the risk of exfoliation of the previously dehydrated epithelial cells of the nose and even their complete separation. Repeated stretching and compression can negatively affect the functionality of the epithelium and, with repeated exposure and damage, lead to structural and functional changes.

Rinsing the nose with a hypertonic or isotonic solution of seawater is a potential solution for nasal obstruction because after rinsing, the airflow through the nose improves and symptoms of obstruction are reduced. However, the effects of using nasal lavage solutions along with exercise in elite athletes are not yet known. The potential synergy of exercise and isotonic seawater solution as a nasal spray on airflow and the subjective impression of nasal patency in healthy individuals has not been sufficiently investigated5.

Research question

What is the effect of an isotonic seawater solution applied as a nasal spray on nasal airflow and the subjective impression of nasal obstruction in healthy athletes?

Hypothesis

An isotonic seawater solution applied as a nasal spray will improve nasal airflow and the subjective impression of nasal obstruction in healthy athletes.

DETAILED DESCRIPTION:
Subjects and Methods

Participants:

50 healthy adult athletes between the ages of 18 and 35 will be engaged in the research (power analysis with 80% power and an alpha error of 5% shows that 32 subjects in two groups are sufficient).

Exclusion criteria: Bacterial or viral acute inflammation of the upper respiratory system, chronic obstruction of one or both nostrils with significant deformation of the septum, surgery on the nose or nasal septum within one month of the start of the study

Isotonic seawater:

product from the market, Aqua Maris nasal spray (manufacturer JGL, Rijeka), applied in accordance with the approved Instructions for Consumers

Study design:

A randomized, interventional prospective cohort study.

Intervention:

The participants will be divided into two groups using the binary coin-toss method (random.org) with similar physical and demographic characteristics. The first group will use an isotonic seawater solution as a nasal spray for 10 days, while the control group will not use such a solution. The group with the isotonic seawater solution applied as a nasal spray will use it at least three times a day, and necessarily before exercise (about 20 minutes before).

Outcome measures:

The primary outcome measures will be nasal airflow measured with a peak nasal inspiratory flow meter (PNIF) and subjective impression of nasal obstruction symptoms before and after exercise by completing the NOSE questionnaire. The NOSE contains five statements about nasal obstruction, divided on a 4-point Likert scale for each statement.

Remark:

PNIF meters will be provided by JGL (measurement with them takes < 1 min/athlete) The NOSE questionnaire (abbreviated from Nasal Obstruction Symptom Evaluation) is an internationally recognized and validated scale for assessing the intensity of nasal obstruction.

The time points for the collection of measures will be:

1. Day 1: before the start of the research, before the first training session (first interval), respectively:

   1. NOSE
   2. PNIF
2. Day 1: after the first use of the spray, (within 20 minutes after the first training session - second interval), i.e. after the first training session in the control group, respectively:

   1. NOSE
   2. PNIF
3. Day 7: after ten days of daily use of the spray, after training (third interval) or after the first training in the control group, respectively:

   1. NOSE
   2. PNIF

Data analysis:

1. Descriptive statistics and inferential statistics will be used to compare outcomes between two groups (no less than 16 participants in the nasal spray group vs. no less than 16 participants without the spray).
2. Each couple from the test group will be joined by a couple from the control group with as similar physical and demographic characteristics as possible.

The Wilcoxon signed rank test and the Friedman test for paired samples will be used depending on the distribution of the data.

Ethical considerations This study will be conducted in accordance with ethical principles and guidelines (1996 Helsinki Declaration, in accordance with current Croatian regulations, and after approval by the competent hospital ethics committee). Written informed consent will be obtained from all participants.

Participants will be informed of the risks and benefits of the study by the examining physician. The confidentiality of the participant's data will be ensured in such a way as to comply with GDPR provisions in accordance with EU and national legislation.

Conclusion

This study aims to investigate the effects of an isotonic solution of seawater from the Adriatic Sea applied as a nasal spray on:

* subjective nasal patency
* nasal airflow in healthy athletes.

The results of this research could help athletes improve performance by improving nasal airflow and nasal function.

ELIGIBILITY:
Inclusion Criteria:

* 50 healthy adult athletes between the ages of 18 and 35 will be engaged in the research (power analysis with 80% power and an alpha error of 5% shows that 32 subjects in two groups are sufficient).

Exclusion Criteria:

* Bacterial or viral acute inflammation of the upper respiratory system, chronic obstruction of one or both nostrils with significant deformation of the septum, surgery on the nose or nasal septum within one month of the start of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak nasal inspiratory flow | Prior to excercise, on the first day after training and on the seventh day after training.
  The primary outcome measures will be nasal airflow measured with a peak nasal inspiratory flow meter (PNIF).
NOSE questionnaire | Prior to excercise, on the first day after training and on the seventh day after training.
  Subjective impression of symptoms of nasal obstruction before and after exercise by completing the NOSE questionnaire. The NOSE contains five statements about nasal obstruction, divided on a 4-point Likert scale for each statement.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No